CLINICAL TRIAL: NCT06089616
Title: An International Observational Registry Study to Further Describe Long-term Safety and Effectiveness of Palovarotene in Patients With Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: A Study to Document and to Further Describe Long-term Safety and Effectiveness of Palovarotene in Participants With Fibrodysplasia Ossificans Progressiva (FOP)
Acronym: FOPal
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60120-453
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fibrodysplasia Ossificans Progressiva
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Cohort: Participants treated with palovarotene (i.e already be receiving palovarotene as prescribed by their treating physician according to locally approved product information)
- Unexposed Cohort: Participants untreated with palovarotene

SUMMARY:
The participants in this registry study will have fibrodysplasia ossificans progressiva (FOP).

FOP is an ultra-rare, severely disabling disease characterized by new bone formation in areas of the body where bone is not normally present (heterotopic ossification (HO)).

HO is often preceded by painful, recurrent episodes of soft tissue swelling (flare-ups).

This registry study will take place in countries where the treatment, known as palovarotene, has been approved for use. Participants will either be treated with palovarotene (i.e already be receiving palovarotene as prescribed by their treating physician according to locally approved product information) or untreated with palovarotene.

The main aim of this registry study will be to collect and assess real-world safety data on children and adult participants with FOP treated with palovarotene.

This registry study will also describe the effectiveness of palovarotene in exposed participants, including the effect on everyday activities and physical performance.

In addition, this registry study aims to descriptively compare key safety outcomes (i.e. flare-up episodes, growth outcomes, and bone fractures) between participants exposed and unexposed to palovarotene.

ELIGIBILITY:
Inclusion Criteria :

* Adult or child with FOP who have been prescribed palovarotene (prior to and independently of the decision to enroll the patient in this registry study and as per local label) by their treating physician according to the locally approved product information;
* Signed informed consent as per local regulations must be obtained and maintained. Consent/assent from the participant should be obtained as appropriate before any registry study data collection are conducted. If applicable, parents or legally authorized representatives must give signed informed consent.

Exclusion Criteria :

* Currently participating in a palovarotene clinical trial;
* Currently participating in any interventional clinical trial for FOP;
* Have any contraindication to palovarotene as per the locally approved label (except for pregnant women who have previously received and discontinued palovarotene at any time during the pregnancy and who will be included for safety follow-up).

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with FOP who have been prescribed palovarotene, as per local label, by their treating physician for which informed consent has been obtained and maintained. Participants cannot be included if they are currently participating in a palovarotene clinical trial or an interventional clinical trial for FOP or if they have any contraindication for palovarotene (except for pregnant women who have previously received and discontinued palovarotene at any time during the pregnancy and who will be included for safety follow-up).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2035-12-05 (Estimated); Study Completion 2035-12-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs), whether or not they are considered as related to palovarotene | From Baseline up to 30 days after the last palovarotene dose.
  Adverse events will be coded according to MedDRA and will be classified by Preferred Term (PT) and system organ class (SOC).
Percentage of Participants With Serious and Non-serious treatment-related TEAEs | From Baseline up to 30 days after the last palovarotene dose.
  Adverse events will be coded according to MedDRA and will be classified by PT and SOC.
Percentage of Participants With all serious TEAEs, whether or not they are considered as related to the palovarotene | From Baseline up to 30 days after the last palovarotene dose.
  Adverse events will be coded according to MedDRA and will be classified by PT and SOC.
Percentage of Participants With nonserious TEAEs whether or not they are considered as related to the palovarotene. | From Baseline up to 30 days after the last palovarotene dose.
  Adverse events will be coded according to MedDRA and will be classified by PT and SOC.

SECONDARY OUTCOMES:
Change from Baseline in Cumulative Analogue Joint Involvement Scale (CAJIS) total score | From Baseline and every six months up to eleven years.
  The CAJIS is an objective measure of joint movement completed by the Investigator to document total joint involvement. The CAJIS total score is calculated as the sum of the scores of all joints/regions and ranges from 0 (no involvement) to 30 (maximally involved).
Change from Baseline in use of assistive devices | From Baseline and every six months up to eleven years.
  Assistive devices is a questionnaire to assess the assistive devices used by particpants and adaptations for their daily living.
Change from Baseline in percent of worst score for Fibrodysplasia Ossificans Progressiva-Physical Function Questionnaire (FOP-PFQ) total score | From Baseline and every six months up to eleven years.
  Fibrodysplasia Ossificans Progressiva-Physical Function Questionnaire (FOP-PFQ) consists of questions which are scored on a scale of 1 to 5, lower scores indicating that the participant has more difficulties.
Change from Baseline in observed and percent predicted Forced Vital Capacity (FVC) | From Baseline and every six months up to eleven years.
  The lung function parameters of observed FVC (liters) and percent predicted FVC are obtained by spirometry.
Change from Baseline in observed and percent predicted Forced Expiratory Volume in one second (FEV1) | From Baseline and every six months up to eleven years.
  The lung function parameters of observed FEV1 (liters) and percent predicted FEV1 are obtained by spirometry.
Change from Baseline in absolute and percent predicted FEV1/FVC ratio | From Baseline and every six months up to eleven years.
  The lung function parameters of the absolute and percent predicted FEV1/FVC ratio are obtained by spirometry.
Change from Baseline in observed and percent predicted Diffusion Capacity of the Lung for Carbon Monoxide (DLCO) | From Baseline and every six months up to eleven years.
  The lung function parameters of observed (traditional unit of mL/min/mmHg or SI unit of mmol/min/kPa) and percent predicted DLCO is obtained by the DLCO test.
Change from Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) physical and mental function (mean global physical and mental health score converted into T-scores) for participants ≥15 years old | From Baseline and every six months up to eleven years.
  PROMIS Global Health Scale for the adult version, the global physical health and global mental health scores will be calculated as follows:
  * Global physical health scores will be calculated as the sum of scores from Questions 3, 6, 7 and 8 and will range from 4 (worse health) to 20 (better health);
  * Global mental health scores will be calculated as the sum of scores from Questions 2, 4, 5 and 10 and will range from 4 (worse health) to 20 (better health).
Change from Baseline in PROMIS overall quality of life (QoL) (mean total score converted into T-scores) for participants <15 years old | From Baseline and every six months up to eleven years.
  PROMIS Global Health Scale for the paediatric version, the total score will be calculated as the sum of scores from the first 7 questions and will range from 7 (worse health) to 35 (better health).
  If more than 3 questions contributing to the total score are missing, the total score will not be calculated. It will be considered as missing.
Change from Baseline in annualized number of Investigator-reported flare-ups by body location and overall | From Baseline and every six months up to eleven years.
  The annualized number of flare-ups will be derived from the number of flare-ups the participant experienced since last visit.
Number of flare-up outcomes | From Baseline and every six months up to eleven years.
  Number of flare-up outcomes as measured by new bone growth, restricted movement at each visit will be reported.
Flare-up Duration | From Baseline and every six months up to eleven years.
  Flare-up duration will be assessed by body location and overall, at each visit.
Number of flare-ups | From 12 months before inclusion Baseline up to eleven years.
Movement mobility change | From Baseline and annually up to eleven years.
  Assessed by key body location: better movement/the same movement/slightly worse movement/moderately worse movement/severely worse movement)
Number of locations impacted per participant | From Baseline and annually up to eleven years.
Evolution of impacted location (how many times a location is impacted) per location | From Baseline and annually up to eleven years.
Movement mobility outcomes: Percentage of participants with new bone growth overall and by flare-up status | From Baseline and every six months up to eleven years.
  The number of extra bone growths, location of the extra bone growth, whether it was preceded by injury, illness, vaccination and/or other events, whether it was preceded by pain, soft tissue swelling, decreased range of motion, stiffness, redness, or warmth, extra bone growth start and stop date and whether it is ongoing, will be collected.
Percentage of participants with any fractures overall | From baseline up to 30 days after the last palovarotene dose.
  Assessed by radiological imaging and clinical examination.
Change from Baseline in annualized number of fractures by body location and overall | From baseline up to 30 days after the last palovarotene dose.
  Assessed by radiological imaging and clinical examination.
Incidence of pregnancy | From Baseline and every month up to 30 days after the last palovarotene dose.
  A pregnant participant with FOP exposed to palovarotene will be followed throughout the pregnancy and the health status of the baby will be verified
Description of pregnancy characteristics and outcomes | From the signing of the ICF and the participant will be followed throughout the pregnancy (From Baseline and every month up to 30 days after the last palovarotene dose) and the health status of the baby will be verified up until one year of age.
  A pregnant participant with FOP exposed to palovarotene will be followed throughout the pregnancy.
Description of pregnancy related Adverse Events (AEs) | From the signing of the ICF and the participant will be followed throughout the pregnancy (From Baseline and every month up to 30 days after the last palovarotene dose) and the health status of the baby will be verified up until one year of age.
  A pregnant participant with FOP exposed to palovarotene will be followed throughout the pregnancy.
Description of birth and developmental outcomes through the first year after birth | From the signing of the ICF and the participant will be followed throughout the pregnancy (From Baseline and every month up to 30 days after the last palovarotene dose) and the health status of the baby will be verified up until one year of age.
  A pregnant participant with FOP exposed to palovarotene will be followed throughout the pregnancy.
Description of birth and developmental outcomes through the first year after birth | From Baseline and every six months up to eleven years.
  Linear height and knee height velocity will be derived for growing children with FOP exposed and unexposed to palovarotene until skeletal maturity or final adult height is reached.
Change from Baseline in height z-score | From Baseline and every six months up to eleven years.
  Linear height z-score will be derived for growing children with FOP exposed and unexposed to palovarotene until skeletal maturity or final adult height is reached.
Mean difference between chronological age and bone age | From Baseline and every six months up to eleven years.
  Bone age (assessment as per the SmPC/PI) and chronological age will be collected for growing children with FOP exposed and unexposed to palovarotene until skeletal maturity or final adult height is reached.
Frequency of premature physeal closure (PPC) overall | From baseline up to 30 days after the last palovarotene dose
  Epiphyseal status ("open" or "closed") (assessment as per the SmPC/PI) will be collected for growing children with FOP exposed and unexposed to palovarotene until skeletal maturity or final adult height is reached.
Mean dose/year of palovarotene for participants with FOP exposed and unexposed to palovarotene for chronic treatment | From Baseline and every six months up to eleven years.
Mean dose/cycle of palovarotene for participants with FOP exposed and unexposed to palovarotene for flare-up treatment | From Baseline and every six months up to eleven years.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (5):
- United States (2):
  - The Regents of the University of California, San Francisco, California
  - The Trustees of the University of Pennsylvania, Office of Clinical Research-Legal Services, Perelman School of Medicine, Philadelphia, Pennsylvania
- Canada (3):
  - Edmonton Clinic Health Academy (ECHA)- University of Alberta, Edmonton
  - Bone Research and Education Centre, Oakville
  - University Health Network (UHN) - Toronto General, Toronto

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/